CLINICAL TRIAL: NCT04322786
Title: The Use of Angiotensin Converting Enzyme Inhibitors and Incident Respiratory Infections, Are They Harmful or Protective? An Analysis Using UK Based Electronic Health Records of 5.6 Million Individuals.
Brief Title: The Use of Angiotensin Converting Enzyme Inhibitors and Incident Respiratory Infections, Are They Harmful or Protective?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: ISAC17_205R
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-03

CONDITIONS: Covid-19, Coronavirus, Angiotensin Converting Enzyme Inhibitors, Influenza, Electronic Health Records, Epidemiology, Comorbidity, Incidence, United Kingdom
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Influenza, Human | interventions — Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACEI user: Individuals with an ACEI prescription in the study population.
  Interventions: Drug: ACE inhibitor
- Matched controls: Individuals without an ACEI prescription, and matched to the users by sex and 10-year age categories.

INTERVENTIONS:
Drug: ACE inhibitor — Any prescription of ACE inhibitor
  Groups: ACEI user

SUMMARY:
The study use UK based linked electronic health records from the Clinical Research Datalink (CALIBER) of 5.6 million individuals to conduct a matched case-control study to investigate the incidence of influenza in individuals prescribed ACEI compared to those not prescribed ACEI.

ELIGIBILITY:
Inclusion Criteria:

* We identify individuals aged 18 years or older and registered in the current primary care practice for at least one year.

Exclusion Criteria:

* We exclude individuals with a prior history of influenza and viral pneumonia before study entry.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The nested case-control study include cases who had an ACEI prescription during study follow-up. We randomly select one control per case from the study cohort of individuals without any documented ACEI use. Controls are matched to incident AF patients according to sex, age (10-year age strata).
Sampling Method: Non-Probability Sample
Enrollment: 1302508 (Actual)
Dates: Start 1998-01-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of influenza | Jan 1st 1998 - May 31st 2016